CLINICAL TRIAL: NCT00727233
Title: Phase I Trial of the Raf Kinase and Receptor Tyrosine Kinase Inhibitor Sorafenib (BAY 43-9006, Nexavar) in Children and Young Adults With Neurofibromatosis Type 1 and Inoperable Plexiform Neurofibromas
Brief Title: Sorafenib to Treat Children and Young Adults With Neurofibromatosis Type 1 and Inoperable Plexiform Neurofibromas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080180; 08-C-0180; NCT01445470 (obsolete NCT alias)
Record Dates: First submitted 2008-07-31; First posted 2008-08-01 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2012-05-04

CONDITIONS: Neurofibromatosis Type I; Plexiform Neurofibroma
Keywords: Neuroblastosis Type I; Plexiform Neurofibromas; Angiogenesis Inhibitor; Kinase Inhibitor; Neurofibromatosis Type 1; NF1; Plexiform Neurofibroma
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform | interventions — Sorafenib; Pharmacokinetics

INTERVENTIONS:
Drug: Nexavar (BAY 43-9006) (Sorafenib)
Drug: Toxicity, Pharmacokinetics
Drug: Pharmacodynamics
Drug: Radiographic Evaluation
Drug: QOL assessment, Neuropsychological
Drug: Bony Toxicity

SUMMARY:
Background:

Patients with neurofibromatosis type 1 are at increased risk of developing tumors called plexiform neurofibromas (PN) that arise from nerves. These tumors are usually non-cancerous, but they can cause serious medical problems.

Sorafenib was recently approved to treat patients with kidney cancer and is now being tested in children with cancer. It affects several pathways thought to be important for the development and growth of PN and may therefore shrink these tumors or slow their growth.

Objectives:

To determine the highest dose of sorafenib that can safely be given to children and young adults with PN.

To identify the side effects of sorafenib in these patients.

To study how the body handles sorafenib by measuring the amount of drug in the bloodstream over time

To determine how the drug affects blood flow and blood cells and proteins.

To determine if sorafenib can shrink or slow the growth of PN.

To determine the effects of sorafenib on learning, attention, memory, and quality of life.

Eligibility:

Patients between 3 and 18 years of age with NF1 who have inoperable PN that can cause significant disability.

Design:

Patients take sorafenib tablets twice a day in 28-day treatment cycles. They may continue treatment until their tumor grows or they develop unacceptable drug side effects. In this dose escalation study, the dosage is increased with every 3 to 6 children who are enrolled until the highest safe dose is determined. In any case, the dose will not exceed that used in children with cancer.

Patients are monitored regularly with physical examinations, blood and urine tests, MRI scans and quality-of-life questionnaires.

Patients whose bones are still growing have periodic x-rays of the hips and lower legs to monitor for possible changes in the structure of growing bones.

Patients have periodic tests of learning and memory before starting treatment and before cycles 4, 12, 18 and 24.

Patients have pharmacokinetic studies to examine how the body handles sorafenib. blood samples are drawn before the first dose of sorafenib and then at 30 minutes, 1 hour, 2 hours, 3 hours, 5 hours, 8 hours, 10 to 12 hours, 24 hours and 30 to 36 hours following the first dose.

...

DETAILED DESCRIPTION:
Background:

* Patients with Neurofibromatosis 1 (NF1) have an increased risk of developing tumors of the central and peripheral nervous system, including plexiform neurofibromas (PN), which are benign nerve sheath tumors that are among the most debilitating complications of NF1. Plexiform neurofibromas may be congenital and appear to have the fastest growth rate in young children. There are no standard treatment options for PN other than surgery, which is often difficult due to the extensive growth and invasion of surrounding tissues.
* Plexiform neurofibromas are composed of neoplastic Schwann cells that lack NF1 gene expression resulting in upregulation of Ras, which initiates several signaling cascades regulating cell proliferation. In addition, PN over express epidermal and platelet derived growth factor receptor and vascular endothelial growth factors, which may promote angiogenesis.
* Sorafenib, a novel orally bioavailable, bi-aryl urea, is a potent inhibitor of raf kinase and a number of receptor tyrosine kinases, which is currently undergoing evaluation in adult cancers, and may mediate anti-tumor effects in PN by several mechanisms.

Objectives:

* To determine the maximum tolerated dose (MTD) of oral sorafenib administered daily to pediatric patients with NF1 and inoperable PN.
* To define the acute and chronic toxicities, pharmacokinetics, and pharmacodynamics of sorafenib.
* To evaluate for potential bone toxicities of sorafenib such as growth plate expansion and growth retardation using automated volumetric MRI analysis of growth plates, multiple measures for height and growth, dual-energy x-ray absorptiometry to evaluate bone mineral density, and laboratory measurements for evaluation of bone turnover and metabolism.
* To determine the effect of sorafenib on the growth rate of PN, quality of life, and cognitive function while on treatment with sorafenib.

Eligibility:

- Pediatric Patients (3-18 years) with NF1 and inoperable measurable PN that have the potential to cause significant morbidity.

Design:

* Sorafenib will be administered orally BID on a continuous dosing schedule (28 days = 1 treatment cycle). Limited dose escalations will be performed to define the MTD based on tolerability of sorafenib during the first three treatment cycles.
* Disease status will be evaluated using volumetric MRI analysis at regular intervals.
* The plasma pharmacokinetics and pharmacodynamics of sorafenib will be evaluated.
* Cognitive function and quality of life outcomes will also be assessed in a pilot fashion to define measures to be used in subsequent phase II trials.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Age: greater than or equal to 3 years and less than or equal to 18 years of age at the time of study enrollment. The upper age limit is in place because early childhood and puberty are considered to be the greatest risk for disease progression, and where sorafenib may have the most benefit. In addition, an important objective of this study is to characterize the pharmacokinetics of sorafenib in the pediatric population since it has been well studied in adults.
2. Diagnosis: Patients with NF1 and inoperable PNs that have the potential to cause significant morbidity, such as (but not limited to) head and neck lesions that could compromise the airway or great vessels, brachial or lumbar plexus lesions that could cause nerve compression and loss of function, lesions that could result in major deformity (e.g., orbital lesions) or significant cosmetic problems, lesions of the extremity that cause limb hypertrophy or loss of function, and painful lesions. Histologic confirmation of tumor is not necessary in the presence of consistent clinical and radiographic findings, but should be considered if malignant degeneration of a PN is clinically suspected.

   A PN is defined as a neurofibroma that has grown along the length of a nerve and may involve multiple fascicles and branches. A spinal PN involves two or more levels with connection between the levels or extending laterally along the nerve. In addition to PN, all study subjects must have either positive genetic testing for NF1 or have at least one other diagnostic criterion for NF1 listed below (NIH Consensus conference:
   * Six or more cafe-au-lait spots (greater than or equal to 0.5cm in prepubertal subjects or greater than or equal to 1.5 cm in post pubertal subjects)
   * Freckling in axilla or groin
   * Optic glioma
   * Two or more Lisch nodules
   * A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
   * A first-degree relative with NF1
3. Measurable disease: Patients must have at least one measurable PN, defined as a lesion of at least 3 cm measured in one dimension. Patients who underwent surgery for resection of a PN are eligible provided the PN was incompletely resected and is measurable as per criteria above.
4. Prior Therapy: Patients with NF1 will only be eligible if complete tumor resection is not feasible, or if a patient with a surgical option refuses surgery.

   * Since there is no standard effective chemotherapy for patients with NF1 and PN, patients may be treated on this trial without having received prior medical therapy directed at their PN.
   * May have received less than or equal to 1 myelosuppressive regimen for PN or other tumor manifestations associated with NF1 such as optic glioma.
   * Patients who have received previous investigational agents or biologic therapy, such as tipifarnib, pirfenidone, Peg-Intron, or other VEGFR inhibitors are eligible for enrollment.
   * Growth factors that support platelet or white cell number or function must not have been administered within the past 7 days.
   * Patients who received prior medical therapy for their PN must have recovered from the toxic effects of all prior therapy before entering this study.
5. Performance status: Patients greater than 10 years of age must have a Karnofsky performance level of greater than or equal to 50%, and children less than or equal to 10 years old must have a Lansky performance of greater than or equal to 50% (Appendix I).
6. Hematologic Function: Patients must have an absolute neutrophil count greater than or equal to 1500/microl, hemoglobin greater than or equal to 9g/dl, and platelet greater than or equal to 100,000/microl.
7. Coagulation: Patients must have adequate hemostatic function defined as PT and PTT less than or equal to 1.5 times ULN. Patients receiving prophylactic anticoagulation for thrombosis are eligible if they meet criteria for adequate hemostatic function (PT and PTT less than or equal to 1.5 times ULN) and thrombotic episode occurred 3 months prior to enrollment. Use of anticoagulants or thrombolytics for care and maintenance of central venous catheters is acceptable.
8. Hepatic Function: Patients must have bilirubin within the upper limit of normal for age, and ALT within the upper limit of normal for age.
9. Serum lipase and amylase within upper limits of normal.
10. Renal Function: Patients must have a creatinine clearance or radioisotope GFR greater than or equal to 60ml/min/1.73 m(2) or a normal serum creatinine based on age described in the table below.

    Age (years) less than or equal to 5 Maximum Serum Creatinine (mg/dL) 0.8

    Age (years) 5 less than or equal to 10 Maximum Serum Creatinine (mg/dL) 1.0

    Age (years) 10 less than or equal to 15 Maximum Serum Creatinine (mg/dL) 1.2

    Age (years) greater than 15 Maximum Serum Creatinine (mg/dL) 1.5
11. Blood pressure: Patients must have a systolic and diastolic blood pressure less than 95th percentile for age and gender (Appendix II) measured as described in section 2.2.
12. Informed Consent: Diagnostic or laboratory studies performed exclusively to determine eligibility for this trial must only be done after obtaining written informed consent from all patients or their legal guardians (if the patient is less than 18 years old). When appropriate, pediatric patients will be included in all discussions. This can be accomplished through one of the following mechanisms: a) the NCI, POB screening protocol, b) an IRB-approved institutional screening protocol or c) the study-specific protocol. Documentation of the informed consent for screening will be maintained in the patient s research chart. Studies or procedures that were performed for clinical indications (not exclusively to determine eligibility) may be used for baseline values even if the studies were done before informed consent was obtained.
13. Durable Power of Attorney (DPA): All patients greater than 18 years of age will be offered the opportunity to assign DPA so that another person can make decisions about their medical care if they become incapacitated or cognitively impaired.

EXCLUSION CRITERIA:

1. Pregnant or breast-feeding females are excluded due to risks of fetal and teratogenic adverse events as seen animal studies. Pregnancy tests must be obtained prior to enrollment on this study in girls, age 9 or older. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method. Abstinence is an acceptable method of birth control.
2. Sorafenib is predominantly metabolized via CYP3A4, and patients who take cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine or Phenobarbital), rifampin, grape fruit, or St. Johns Wort will not be eligible for the trial. Patients must have discontinued these medications at least 7 days prior to enrollment of trial.
3. Patients who have had major surgery within the past 3 months are excluded. Patients having minor surgery (i.e., central line placement) within the past 2 weeks are excluded.
4. An investigational agent within the past 30 days.
5. Ongoing radiation therapy, chemotherapy, hormonal therapy directed at the tumor, immunotherapy, or biologic therapy.
6. Clinically significant uncontrolled unrelated systemic illness such as serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction.
7. Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
8. Inability to swallow tablets, since tablets cannot be crushed or broken.
9. Inability to undergo MRI and/or contraindication for MRI examinations following the MRI protocol (Appendix III). Prosthesis or orthopedic or dental braces that would interfere with volumetric analysis of target PN on MRI.
10. Prior treatment with sorafenib.
11. Evidence of an optic glioma, malignant glioma, malignant peripheral nerve sheath tumor, or other cancer requiring treatment with chemotherapy or radiation therapy.
12. Patients with a history of arterial or venous thrombosis with in the prior 3 months.
13. Patients who experienced significant hemorrhage (hemoptysis, melena, or hematemesis) within the past 2 weeks or with a history of bleeding diathesis.
14. Patients with a history of NF1 related cerebral vascular anomaly.
15. Patients requiring systemic full dose anticoagulation with systemic thrombolytics, heparin, coumadin, or low molecular weight heparin or other anticoagulants for therapy of active thrombosis within the prior 3 months.
16. Patients on anti-hypertensive medications and patients with baseline hypertension (greater than or equal to 95th % for age and gender, see Appendix II) (treated or untreated).

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2008-07-08; Primary Completion 2011-06-16 (Actual); Study Completion 2011-06-16 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose, chronic toxicity, pharmacokinetics and pharmacodynamics.

SECONDARY OUTCOMES:
3D MRI of plexiform neurofibromas, pharmacodynamics, cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Widemann BC, Salzer WL, Arceci RJ, Blaney SM, Fox E, End D, Gillespie A, Whitcomb P, Palumbo JS, Pitney A, Jayaprakash N, Zannikos P, Balis FM. Phase I trial and pharmacokinetic study of the farnesyltransferase inhibitor tipifarnib in children with refractory solid tumors or neurofibromatosis type I and plexiform neurofibromas. J Clin Oncol. 2006 Jan 20;24(3):507-16. doi: 10.1200/JCO.2005.03.8638. PMID 16421428
- [Background] Korf BR. Plexiform neurofibromas. Am J Med Genet. 1999 Mar 26;89(1):31-7. doi: 10.1002/(sici)1096-8628(19990326)89:13.0.co;2-w. PMID 10469434
- [Background] Friedman JM. Neurofibromatosis 1: clinical manifestations and diagnostic criteria. J Child Neurol. 2002 Aug;17(8):548-54; discussion 571-2, 646-51. doi: 10.1177/088307380201700802. PMID 12403552